CLINICAL TRIAL: NCT02379130
Title: FNI Between Mothers and Preschool Age Children
Brief Title: Early Behavioral Intervention for Preterm Infants
Acronym: EBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment/retention
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G. Welch, MD, Associate Professor of Psychiatry in Pediatrics and Pathology and Cell Biology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AAAO2957
Record Dates: First submitted 2015-02-25; First posted 2015-03-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Premature Birth
Keywords: Premature; Family Nurture Intervention
MeSH Terms: conditions — Premature Birth | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Nurture Intervention Group (Experimental): Children in the FNI group will continue to attend any intervention programs that they are already enrolled in. In addition, they will be asked to attend 1 clinic visit per week for 6 weeks over the course of 12 weeks. During each visit, the mother-child will meet with trained Nurture Specialists. The Nurture Specialists will facilitate and encourage the mother and child to engage in nurturing and calming activities, including sustained touch, vocal soothing, and an odor cloth exchange. FNI families will be asked to participate in a 6 month post-enrollment follow-up visit and a 12 month post-enrollment follow-up visit.
  Interventions: Behavioral: Family Nurture Intervention
- Play and Nutrition Intervention Group (Active Comparator): Children in the PNI group will continue to attend any intervention programs that they are already enrolled in. They will be asked to attend 1 clinic visit per week for 6 weeks over the course of 12 weeks to meet with clinical personnel who will collect measures regarding the child's behavior and development. At each visit, study staff will meet with mothers to facilitate a lesson plan on appropriate play and nutrition. NPI families will be asked to participate in a 6 month post-enrollment follow-up visit and a 12 month post-enrollment follow-up visit.
  Interventions: Behavioral: Play and Nutrition Intervention

INTERVENTIONS:
Behavioral: Family Nurture Intervention — The intervention begins with Block play. The child will be asked to play blocks with the mother during a eight minute video acquisition which will be coded for mother child interaction analysis. At the end of the video period the child will sit on the mother's lap. The pair will be asked to talk and play with each other as they customarily do. If the child becomes restless the mother will be coached by the nurture specialist to further engage the child with soothing and calming; the mother will be helped to bring the child back into a calm state through sustained physical contact, comfort touch, soothing words, and eye contact. The mother will also be helped to verbally express her feelings toward her child and to tolerate her child's full range of feeling.
  Other Names: FNI
  Arms: Family Nurture Intervention Group
Behavioral: Play and Nutrition Intervention — The intervention begins with Block play. The child will be asked to play blocks with the mother during a eight minute video acquisition which will be coded for mother child interaction analysis. At the end of the video period, the child and mother will play nutrition-focused games using the Healthy Habits for Life program designed by Michelle Obama.
  Other Names: PNI
  Arms: Play and Nutrition Intervention Group

SUMMARY:
The purpose of this study is to determine the effects of Family Nurture Intervention in preschool aged children between 2.5 and 4.5 years of age who were born prematurely and exhibit developmental deficits. The new approach is based on improving aspects of maternal nurturing behaviors as well as mother-child co-regulation, which are important to early development. Since young children with developmental deficits are often easily upset, mothers will be taught how to co-regulate with their child through comfort and calming interactions during 11 clinic visits. Assessments in the follow-up clinic will test the immediate and long-term effects of this new approach to the nurture of children who were born early and demonstrate developmental problems and behavioral problems.

DETAILED DESCRIPTION:
Mother-infant interactions are the foundation for the organization of the infant's neurobiological, sensory, perceptual, emotional, physical, and relational systems (Hofer, 1987). For the developing infant, one of the most critical sources of regulatory input is through contact with the mother and her nurturing behavior. The infant's responses to the mother provide feedback that shapes her behavior as well. There are many co-regulatory processes embedded in these synchronous and reciprocal interactions which cross neurophysiological and neurobehavioral domains (Als, 1999). A necessary but detrimental separation between mother and infant is created at a critical period when mother-infant co-regulation should be developing. Regardless of NICU or well-baby nursery care, the physiological challenges associated with being born too soon, along with disturbances in normal mother-infant interactions are key factors underlying the risks of early and late preterm infants for a broad range of early and midlife disorders (DeBoer, et al., 1984 if this does not include late preterm, find another reference). This study compares common early interventions such as occupational, physical, and speech therapy with a Family Nurture Intervention (FNI), instituted at age 3 to 4 for preschool aged children with developmental delays. This is a developmental time point at which delays including deficits in emotion regulation, language, cognition, and attention are identifiable. The investigators hypothesize that the Family Nurture Intervention will alter a wide range of physiological regulatory capacities and will result in improved indices of mother psychological and child neurobehavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infant is a singleton (matched between groups)
* Mother is 18 years of age or older
* Mother has at least one supporting person in the home (e.g. significant other, mother, father, sibling, aunt, grandmother, step-parent)
* Child demonstrates developmental deficit (language, cognition, motor, emotion)

Exclusion Criteria:

* The child has severe congenital anomalies including chromosomal anomalies
* The child has severe motor or physical disability
* Mother currently presents with psychosis or is currently taking antipsychotic medication
* Status of enrolled subject changes and subject no longer falls in inclusion criteria
* Mother and/or infant has a medical condition that precludes intervention components
* Mother and/or infant has a contagion that endangers other participants in the study

Ages: 30 Months to 40 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Child Behavior Checklist (CBCL) Scale | Baseline, 5 weeks, 6 months, 12 months
  The Child Behavior Checklist (CBCL) is a device by which parents rate a child's problem behaviors and competencies. The CBCL can also be used to measure a child's change in behavior over time or following a treatment. The CBCL consists of 100 items.

SECONDARY OUTCOMES:
Salivary Cortisol Level | Up to 3 years
  Cortisol is the hormone produced at the end of the Hypothalamic-Pituitary-Adrenal (HPA) Axis and is used to measure stress levels. Mothers and children will be asked for a saliva sample for cortisol determination throughout the intervention program.
Oxytocin (OT) Level | Up to 3 years
  In this study OT will be measured in urine and saliva of both mother and child to determine the extent to which OT is different in control and intervention subjects. Release of OT under conditions of isolation/stress may help protect mammals against the effects of stress.
Variance in Vagal Tone (High Frequency Heart Period Variability) | Up to 3 years
  Using data obtained during each follow-up visit, we will characterize various parameters of cardiac function and regulation including assessments of parasympathetic modulation of heart rate.Heart rate and respiration will be digitized at 2000 samples/sec, and undergo further mean and interval calculations.
Strengths and Difficulties Questionnaire (SDQ) Score | Up to 3 years
  SDQ is a brief parent-report behavioral screening questionnaire for 3-16 year olds. It consists of 25 items that are divided into 5 categories: emotional problems, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.
Sleep Habits Questionnaire (SHQ) Score | Up to 3 years
  SHQ is a 64-item parent report instrument about their child's sleep across the first 5 years of life, beginning at age 6 months.
State-Trait Anxiety Inventory (STAI) Scale | Up to 3 years
  STAI is the definitive instrument for measuring anxiety. It comprises 2 separate self-report scales of 20 items each that measure state and trait anxiety (Spanish version also available). The S-Anxiety Scale (measuring state), has been found to be a sensitive indicator of changes in transitory anxiety. The T-Anxiety scale has proven useful for identifying persons who differ in motivation or drive level. The STAI has been used in studies examining parents of hospitalized children, the transition to a maternal role, and perception of illness severity in infants.
Parenting Stress Index (PSI) Scale | Up to 3 years
  We will be using the short form of 36 items, which only requires 10 mins to complete. This form of the PSI (1983) is from a 101 item questionnaire that includes the following 13 scales: Adaptability, Acceptability, Demandingness, Mood, Distractibility/Hyperactivity, Reinforces Parent, Depression, Attachment, Restriction of Role, Sense of Competence, Social Isolation, Relationship with Spouse, and Parent Health.
Center for Epidemiologic Studies Depression (CES-D) Score | Up to 3 years
  The CES-D is a 20 item self-report inventory designed to assess current but nonspecific distress rather than clinically diagnosed depression. Criteria are based on DSM-IV criteria for depressive disorders. A score of 16+ is traditionally used to select a depressed group.
Maternal Self Efficacy Scale | Up to 3 years
  This is a 10 item measure designed to measure feelings of efficacy in mothers of infants aged 3 to 131 months. Mothers rate their perceived efficacy across a variety of childcare activities along a 4-point scale.
Norbeck Social Support Questionnaire (NSSQ) Score | Up to 3 years
  Respondents are asked to list first names or initials for each significant person in their lives who provides personal support to them. Then they indicate the kind of relationship for each person on this network list. Using a 5-point rating scale they describe the amount of support available from each person on their network list for 8 questions.
Mom's Support Circle Scale | Up to 3 years
  This questionnaire was specifically created for the current study. It assesses who will support and who is supporting the mom with her child. It assess how 'available' and 'helpful' each potential support person (e.g., husband, sibling, grandparent, friend) is on a rating scale from rated from 1 (less) to 5 (more).

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Ludwig, BA, Study Director — Lab Manager, Nurture Science Progam, Columbia University Medical Center; Martha G Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - Nuture Science Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided